CLINICAL TRIAL: NCT07219342
Title: The Purpose of This Research Study is to Compare the Effectiveness of a Non-fluoride Whitening Toothpaste (Test) to That of a Non-whitening Fluoride Toothpaste (Negative Control) in Improving Tooth Whiteness (Removal of Extrinsic Stains) Over 8 Weeks of Unsupervised Use.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boka LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KOBA-WHT-2025-01
Record Dates: First submitted 2025-09-24; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Teeth Staining
MeSH Terms: conditions — Tooth Discoloration | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whitening Toothpaste (Experimental)
  Interventions: Other: Toothpaste
- Non-Whitening Toothpaste (Placebo Comparator)
  Interventions: Other: Toothpaste

INTERVENTIONS:
Other: Toothpaste — Toothpaste with stain removing abilities

SUMMARY:
The Purpose of This Research Study is to Compare the Effectiveness of a Non-fluoride Whitening Toothpaste (Test) to That of a Non-whitening Fluoride Toothpaste (Negative Control) in Improving Tooth Whiteness (Removal of Extrinsic Stains) Over 8 Weeks of Unsupervised Use.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 65, ambulatory, and in good general health as determined by the Study Examiner, based upon clinical observation and the Medical/Dental History.
* Be able to understand and sign the Informed Consent, complete a Medical History form, understand and comply with al study directions, and be available for al exam periods.
* Present with adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect) and continue to meet the inclusion criteria and not fall into the categories of exclusion during the period of the study.
* Have a mean Macpherson Modified Lobene Stain Index (MLSI) score of ≥ 1.5 on the labial surfaces of at least 8 of 12 anterior teeth.
* Have a minimum of 16 natural teeth, including the four maxillary incisors.
* Have had dental prophylaxis within the past 18 months, but not within the past 3 months, and agree ot refrain from using al oral care products (other dentifrices and toothbrushes, dental floss and mouthwashes), other than their assigned product, for the duration of the study.
* Agree to refrain from using all whitening products and procedures for the duration of the study.
* Drink tea/coffee daily.

Exclusion Criteria:

* Have a history of serious medical conditions or transmittable diseases including but not limited to active hepatitis, heart irregularities, conditions requiring pre-medication for dental procedures, rheumatic heart disease, untreated diabetes mellitus, cirrhosis, leukemia, phenylketonuria, renal disease, sarcoidosis, tuberculosis, bleeding disorder, vascular disease, AIDS, history of drug allergies or idiosyncrasies, or any other medical condition that may preclude successful participation ni the trial, at the discretion of the Study Examiner.
* Have had prior significant adverse effects following the use of oral hygiene products.
* Have the presence of orthodontic bands, retainers, fixed appliances, large restorations, or removable partial dentures, which may interfere with clinical assessments of the evaluable teeth.
* Show evidence of neglected dental health in need of prompt professional attention (i.e., gross calculus deposits or rampant caries), significant oral soft tissue pathology, systemically related gingival enlargement, generalized recession, tissue damage due to ill-fitting appliances or restorations, or extreme crowding or overlapping of teeth. Periodontitis (ADA Class I, III, or IV), e.g., more than two teeth with periodontal pockets >4 mm as evidenced by purulent exudate, tooth mobility, and other signs indicating that the integrity of the data collected might be compromised.
* Have medication therapy that is current and ongoing or within the past 4 weeks, which might interfere with the outcome of the study by affecting oral tissue condition, salivation, or stain formation (particularly chronic long-term medication therapy).
* Are nursing (breast-feeding) or pregnant.
* Present at baseline with any reported sensory reactions, observed gum irritation, or any condition that would interfere with subsequent clinical assessments, or subjects with a history of allergy to oral care products, severe oral cavity sensitivity, or excessive oral irritation.
* Have participated in tooth bleaching or whitening dentifrice trials within the last three months.
* Have had professional or at-home bleaching during the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-11-06 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Tooth color | 8 weeks
  The Modified Lobene Stain Index (MLSI) Area x Intensity score for the overall tooth surfaces will be used for measurment of tooth color.
  The Primary Endpoint is the MLSI (extrinsic stain mean scores) at the 8-week timepoint compared to baseline. The between treatments would also be a primary endpoint after 8 weeks of unsupervised use.

SECONDARY OUTCOMES:
Whitening | 8 Weeks
  To determine the improvement in tooth shade as measured by Classic Vita Shade Guide after 8 weeks of use of the two dentifrices as compared to their respective baseline shades.
  The Secondary Endpoint is the L*a*b* comparison after 8 weeks of use, both within and between treatment groups. Classic Vita Shade Guide.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, DDS, MPA, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No